CLINICAL TRIAL: NCT04485299
Title: Quantitative Clinical Assessment of Bifluorid 10 Versus Varnish Fluoride on The Exposed Hypersensitive Cervical Dentin in Adult Patient: A Randomized Clinical Trial
Brief Title: Clinical Assessment of Bifluorid 10 vs Varnish Fluoride on The Exposed Hypersensitive Cervical Dentin in Adult Patient
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zaid Yousef Fakhry Al khateeb, Master's degree student - faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPR 20/7/2020
Record Dates: First submitted 2020-07-19; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Hypersensitivity; Dentin Sensitivity
MeSH Terms: conditions — Hypersensitivity; Dentin Sensitivity | interventions — Sodium Fluoride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- bifluorid 10 varnish (Experimental): Bifluorid 10 (NaF and CaF) lead to reduce the dentin hypersensitivity, the sodium fluoride (NaF) dissociates and releases F ions, that diffuse through the tubules and then precipitates as calcium fluoride as a consequence of the high of calcium content in saliva and dentinal fluid ,The calcium fluoride (CaF) present in the varnish composition diffuses into the tubules and block the canal with a semi-permanent protective layer.The calcium fluoride is added to block the dentin tubules mechanically, by the combination with the calcium fluoride resulted from the sodium fluoride reaction to the calcium of dentin.
  Interventions: Drug: Bifluorid 10 ,VOCO
- sodium fluoride varnish (Active Comparator): Topical application of varnish fluoride (sodium fluoride NaF) effect on exposed dentine as a desensitizing agent, the varnish fluoride process is caused by the reaction between NaF and calcium ions resulting in calcium fluoride crystals being deposited on the openings of the dentinal tubules that decrease pain.
  Interventions: Drug: Sodium Fluoride 5% Dental Varnish

INTERVENTIONS:
Drug: Bifluorid 10 ,VOCO — NaF and CaF 10 %
  Other Names: Bifluorid 10
  Arms: bifluorid 10 varnish
Drug: Sodium Fluoride 5% Dental Varnish — 5% NaF
  Other Names: conventional sodium fluoride varnish
  Arms: sodium fluoride varnish

SUMMARY:
Aim of the study will be conducted to compare the efficacy of bifluoride (NaF and CaF) versus conventional fluoride varnish (Sodium Flouride) in the management of hypersensitivity of exposed cervical area in adult patients over 2 month

ELIGIBILITY:
Inclusion Criteria:

* Healthy patient with free medical history.
* Age range 18-60 years old.
* Good oral hygiene
* Patients suffering from pain due to dentin hypersensitivity.
* Patient with sound first molar .

Exclusion Criteria:

* Patients using desensitizing agents, receiving periodontal treatment or had received nonsurgical periodontal treatment in the last three months.
* Patient wearing orthodontic appliance.
* Patient with teeth having a painful condition involving the pulp and periapical region.
* Patients who had allergy to materials will be used in the study.
* Pregnancy.
* Patient who does not consent to participation.
* Patient who does not attend to the follow up.
* A patient who has a carious first molar.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Dentin hypersensitivity | pre-intervention
  measurement of dentin hypersensitivity by VAS scale
Dentin hypersensitivity | 2 min
  measurement of dentin hypersensitivity by VAS scale
Dentin hypersensitivity | 1 week
  measurement of dentin hypersensitivity by VAS scale
Dentin hypersensitivity | 4 weeks
  measurement of dentin hypersensitivity by VAS scale
Dentin hypersensitivity | 8 weeks
  measurement of dentin hypersensitivity by VAS scale

SECONDARY OUTCOMES:
Dentinal tubule occlusion | Pre-intervention
  Percentage of dentinal tubule occlusion measure by scanning electron microscope SEM
Dentinal tubule occlusion | 8 weeks
  Percentage of dentinal tubule occlusion measure by scanning electron microscope SEM